CLINICAL TRIAL: NCT04501484
Title: Bilateral Essential Tremor Treatment With Magnetic Resonance-guided Focused Ultrasound
Brief Title: Bilateral Essential Tremor Treatment With FUS
Acronym: BEST-FUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-5172
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Essential Tremor
Keywords: High-Intensity Focused Ultrasound Ablation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Masking Description: All assessments filmed on video and scored by a blinded evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Participants will undergo a thalamotomy contralateral to their previous treatment with MRgFUS using ExAblate Neuro 4000 device (InSightec Ltd, Tirat Carmel, Israel).
  Interventions: Procedure: Magnetic Resonance-guided Focused Ultrasound VIM Thalamotomy

INTERVENTIONS:
Procedure: Magnetic Resonance-guided Focused Ultrasound VIM Thalamotomy — Ablation of contralateral VIM nucleus of thalamus with MRgFUS using ExAblate Neuro 4000 Device (InSightec Ltd, Tirat Carmel, Israel)

SUMMARY:
Combined Phase II/III, multi-center, prospective, single-blinded trial.

Ten (10) patients with who previously underwent successful and uncomplicated MRgFUS thalamotomy for essential tremor will undergo a contralateral treatment. The incidence of side effects will be determined at 1 and 3 months postoperatively, graded per the CTCAE v5 and analyzed by a data safety monitoring board. Upon successful review, this Phase II trial will be converted to a Phase III trial of utility that will enrol 40 additional patients. The primary outcome will be the change in QUEST score at 12 months postoperatively, as well as a patient-reported assessment of Health Utility. Secondary outcomes will include objective tremor, gait and speech assessments (filmed and scored by blinded evaluators), as well as quality of life questionnaires and adverse events questionnaires. Outcomes will be assessed immediately after the procedure, as well as 1, 3, 12, 24 and 36 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years
* The patient has a primary diagnosis of ET or ET plus confirmed by a movement disorder neurologist;
* The patient previously underwent a MRgFUS (> 6 months ago);
* The tremor on the untreated side negatively impacts the patients' quality of life;
* The patient wants treatment of the contralateral side.

Exclusion Criteria:

* Clinically relevant gait and/or balance impairment (e.g. wide-based, more than 2 falls/months, wheelchair, walker, cane use)
* Clinically relevant speech impairment (e.g. impairment of intelligibility)
* Inability to comply with the follow-up schedule;
* Refusal of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in QUEST Score | 12 months
  Difference in QUEST score between baseline and the 12-month follow-up, with statistical significance defined as p = 0.05 and a minimum clinically important difference (MCID) defined as 5
Patient-based Assessment of Utility | 12 months
  A patient-reported assessment of utility after 12 months using the question "Knowing what you know now, would you do this treatment again?".

SECONDARY OUTCOMES:
Gait Assessment (NRS-11) | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Patient-reported and blinded observer rating of the patient's ability to walk (Numerical rating scale (NRS-11) from 0 to 10, with 10 being best)
Gait Assessment (missteps) | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Number of missteps in a 6 m standardized tandem walk
Falls | Post operative month 1, 3, 12, 24, 36
  Number of falls in last month
Speech Assessment (NRS-11) | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Patient-reported and blinded observer rating of the patient's ability to speak (Numerical rating scale (NRS-11) from 0 to 10, with 10 being best)
Numbness | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Incidence of new-onset numbness
Dysgeusia | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Incidence of taste alterations
Other adverse events | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Incidence of other adverse events as classified in the CTCAE
Tremor (CRST) | Immediately after surgery, post operative month 1, 3, 12, 24, 36
  Assessment of tremor using the Clinical Rating Scale for Tremor (CRST) parts A (0-88) and B (0-36), higher scores correspond to a worse tremor).
Quality of life (QUEST) | Post operative month 1, 3, 12, 24, 36
  QUality of life in ESsential Tremor (QUEST) questionnaire (0-100%, higher scores correspond to a worse quality of life)
Quality of life (CRST part C) | Post operative month 1, 3, 12, 24, 36
  Part C of the Clinical Rating Scale for Tremor (CRST) (0-32, higher scores correspond to a worse quality of life)
Health Utility (EQ-5D-5L) | Post operative month 1, 3, 12, 24, 36
  Health Utility measured using the EQ-5D-5L and computed using the Canadian preference weights. Values range from 0 to 1, with 1 representing a perfect health.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lozano, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No